CLINICAL TRIAL: NCT04447183
Title: A Phase II Study of the Safety and Effectiveness of rhTSH in Radioiodine Treatment for Patients With Differentiated Thyroid Cancer.
Brief Title: The Safety and Effectiveness of rhTSH in Radioiodine Treatment for Patients With Differentiated Thyroid Cancer.
Acronym: DTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGTSH002
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — Thyrotropin Alfa; Injections

STUDY DESIGN:
Intervention Model Description: A randomized, open, parallel controlled, multi-center clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test group of patients who took thyroid hormone medicine and were euthyroid [i.e. their thyroid stimulating hormone (TSH) levels are normal], and received injections of Thyrogen (0.9 mg daily on two consecutive days) followed by oral radioiodine.
  Interventions: Drug: Recombinant Human Thyroid Stimulating Hormone for Injection(rhTSH); Other: radioactive iodine
- Control group (Experimental): The control group of patients did not take thyroid hormone medicine so that they were hypothyroid (i.e. their TSH levels were high,TSH≥30mU/L), and were given oral radioiodine.
  Interventions: Other: radioactive iodine

INTERVENTIONS:
Drug: Recombinant Human Thyroid Stimulating Hormone for Injection(rhTSH) — rhTSH: 0.9 mg IM daily on two consecutive days;radioactive iodine: 30mCi±1.5mCi or 1.11GBq of 131I oral
  Other Names: radioactive iodine
  Arms: Test group
Other: radioactive iodine — radioactive iodine: 30mCi±1.5mCi or 1.11GBq of 131I oral

SUMMARY:
This is a randomized, open, parallel controlled, multi-center clinical trial; 120 subjects were randomly assigned to the test group and the control group according to 3:1.

DETAILED DESCRIPTION:
This study was conducted in patients with differentiated thyroid cancer who had undergone near-total thyroidectomy. After surgery patients were randomized to one of two methods of performing thyroid remnant ablation (use of radioiodine to remove any remaining thyroid tissue). One group of patients who took thyroid hormone medicine and were euthyroid [i.e. their thyroid stimulating hormone (TSH) levels are normal], and received injections of Thyrogen (0.9 mg daily on two consecutive days) followed by oral radioiodine. The second group of patients did not take thyroid hormone medicine so that they were hypothyroid (i.e. their TSH levels were high), and were given oral radioiodine. All patients received the same amount of radioactive iodine (30mCi±1.5mCi or 1.11GBq of 131I). Approximately 9 months later, whole body scans were performed on all patients to learn whether the thyroid remnants had been successfully ablated.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of differentiated thyroid cancer, including papillary thyroid cancer (including papillary carcinoma follicular subtype), follicular thyroid cancer, and Hurthle cell thyroid cancer;
* Patients who were at 18~75 years old (male or female).
* Patients with a total or near-total thyroidectomy within 12 weeks prior to enrollment and plan to performing radioactive iodine((131)Ⅰ) thyroid remnant ablation.
* Serum TSH ≤ 0.5 mU/L；
* Women of childbearing age are HCG-negative;
* Low iodine diet before enrollment for more than 4 weeks;
* Patients are voluntarily enrolled, and written informed consent forms can be used for treatment and visits as required by the program.

Exclusion Criteria:

* Any significant clinical and laboratory abnormalities (eg, severe cardiopulmonary disease, hepatic insufficiency, renal function Incomplete, congestive heart failure, advanced lung disease or advanced cardiovascular and cerebrovascular disease, active infection);
* Patients who have used any water-soluble radiographic contrast agent intravenously, underwent intrathecal iodine angiography or gallbladder iodine imaging within 3 months before administration;
* Taken/eaten within 4 weeks prior to administration Drugs/foods that affect iodine uptake or metabolism, such as multivitamins, glucocorticoids, diuretics, lithium, thiouracil, tazobactam, algae, iodine (except thyroid hormone replacement therapy);
* Before administration Stroke, unstable angina (CCS class II or higher), atrial fibrillation or medication (within beta blocker or digoxin) within 6 months Patients with a history of arrhythmia;
* Pregnant or lactating women;
* Patients who are allergic to rhTSH and its excipients;
* Patients with positive infection-related tests : Includes hepatitis C、syphilis and AIDS;
* Participated in any drug or medical device clinical trial within 1 month prior to the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Ablation success rate by Diagnostic Whole Body Scan (DxWBS) | at week 36
  In the THW state (TSH≥30mU/L), DxWBS showed the proportion of subjects who did not see radioactive iodine uptake in the thyroid gland.

SECONDARY OUTCOMES:
Serum thyroglobulin (Tg) levels | at week 36
  In the THW state (TSH≥30mU/L), the proportion of patients with Tg levels <1ng/mL and neck B-ultrasound negative during rhTSH stimulation accounted for all subjects.
Adverse Event | up to week 40 ± 7 day
  Classification and degree of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No